CLINICAL TRIAL: NCT06048510
Title: New Markers of Glycation to Predict Gestational Diabetes Mellitus and Macrosomia.
Acronym: GLYCAGEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Société Francophone du Diabète (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/26
Record Dates: First submitted 2023-07-17; First posted 2023-09-21 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Macrosomia, Fetal; Gestational Diabetes Mellitus in Pregnancy
Keywords: skin autofluorescence; glycated albumin,; HbA1c; glycation biomarkers; macrosomia; gestational diabetes mellitus
MeSH Terms: conditions — Fetal Macrosomia; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental): Pregnant women, with gestational age at inclusion <28 weeks of amenorrhea, with or without risk factors for GDM will be included in the first consultation at the Maternity Hospital (Bordeaux University Hospital).
  Determination of glycation markers (HbA1c, glycated albumin, and skin autofluorescence).
  Interventions: Diagnostic Test: Pregnant women

INTERVENTIONS:
Diagnostic Test: Pregnant women — Gestational Diabetes Mellitus increases the risk of adverse pregnancy outcomes (such as macrosomia).
  The lack of early clinical symptoms leads to screen pregnant women for GDM, and the strategies of screening are a matter of debate.
  Interventions to control glucose levels in women with GDM have demonstrated efficacy in terms of macrosomia. However, macrosomia may start before the time of screening, suggesting that markers of glycation may have interest : skin autofluorescence, glycated albumin.

SUMMARY:
Gestational diabetes mellitus (GDM) increases the risk of macrosomia and other adverse pregnancy outcomes. Screening strategies are debated: universal vs. selective, and macrosomia may begin before the time of screening, suggesting that glycation markers may have an interest. The objective of this trail is to compare novel markers: skin autofluorescence and glycated albumin, to HbA1c (reference) as predictors of GDM, macrosomia and other adverse outcomes, in pregnant women.

ELIGIBILITY:
Inclusion criteria:

1. Age ≥ 18 years
2. Singleton pregnancy (or twin pregnancy reduced spontaneously or medically before 14 weeks of amenorrhea)
3. Gestational age at inclusion <28 weeks of amenorrhea
4. Participant affiliated with or beneficiary of a social security scheme
5. Collection of patient consent.

Exclusion criteria:

1. Gestational age at inclusion ≥ 28 weeks of amenorrhea
2. Multiple pregnancy
3. Known diabetes prior to pregnancy
4. History of bariatric surgery
5. Expected delivery in another maternity unit not participating in the study
6. Person deprived of liberty by judicial or administrative decision
7. Guardianship or curatorship
8. Participant not affiliated or not benefiting from a social security scheme.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of GDM diagnosed during pregnancy. | At trimester 1
  The primary outcome is the incidence of GDM diagnosed during pregnancy after inclusion in the trial. The measure is performed by fasting blood glucose:≥ 0.92 g/L and < 1.26 g/L,or based on the result of the 75g OGTT performed at 24-28 weeks of amenorrhea, if glycemia at time 0 ≥ 92 mg/dL (5.06 mmol/L) and/or time 60min ≥ 180 mg/dL (9.9 mmol/L) and/or time 120min ≥153 mg/dL (8.42 mmol/L).

SECONDARY OUTCOMES:
Fetal morbidity | Between the day of delivery and the following day
  Incidence of fetal death in utero
Obstetrical outcome | Between the day of delivery and the following day
  Incidence of labor induction, caesarean section, instrumental delivery.
Maternal morbidity | Between the day of delivery and the following day
  Documentation of maternal morbidity diagnosis
Neonatal morbidity 1 | Between the day of delivery and the following day
  Incidence of macrosomia (by birth weight ≥ 4,000g and Large for Gestational Age if ≥ 90th centiles according to sex and gestational age)
Neonatal morbidity 2 | Between the day of delivery and the following day
  Documentation of neonatal morbidity diagnosis
Neonatal morbidity 3 | Between the day of delivery and the following day
  Hospitalization in neonatology or neonatal intensive care unit
Neonatal morbidity 4 | Between the day of delivery and the following day
  Presence of anoxic-ischemic encephalopath or neonatal seizure

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pellegrin, Bordeaux, France